CLINICAL TRIAL: NCT04981067
Title: Median Effective Concentration of Ropivacaine for Ultrasound-guided Popliteal Sciatic Nerve Block in Patients Undergoing Diabetic Foot Surgery
Brief Title: Dose-finding Study: Popliteal Sciatic Nerve Block in Patients Undergoing Diabetic Foot Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seokha Yoo, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2102-120-1220
Record Dates: First submitted 2021-06-28; First posted 2021-07-28 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot; Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies | interventions — S-Adenosylmethionine

STUDY DESIGN:
Intervention Model Description: The biased coin design up-and-down method
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sciatic nerve block using same or decreased concentration of local anesthetic (Other): If the sciatic nerve block in the previous participant was successful, the concentration of local anesthetic would be maintained or decreased 0.05% in the next patient based on a random assignment.
  Interventions: Other: Maintain the concentration of ropivacaine as same as those used in the previous participant; Other: Decrease the ropivacaine concentration by 0.05% from the concentration used in the previous participant
- Sciatic nerve block using increased concentration of local anesthetic (Other): If the sciatic nerve block in the previous participant was not successful, the concentration of local anesthetic would be increased 0.05% in the next patient.
  Interventions: Other: Increase the ropivacaine concentration by 0.05% from the concentration used in the previous participant

INTERVENTIONS:
Other: Maintain the concentration of ropivacaine as same as those used in the previous participant — Maintain the same concentration of ropivacaine used in the previous participant with an 89% chance through a random assignment
  Arms: Sciatic nerve block using same or decreased concentration of local anesthetic
Other: Decrease the ropivacaine concentration by 0.05% from the concentration used in the previous participant — Decrease ropivacaine concentration by 0.05% from the concentration used in the previous participant with an 11% chance through a random assignment
  Arms: Sciatic nerve block using same or decreased concentration of local anesthetic
Other: Increase the ropivacaine concentration by 0.05% from the concentration used in the previous participant — Increase ropivacaine concentration by 0.05% from the concentration used in the previous participant.
  Arms: Sciatic nerve block using increased concentration of local anesthetic

SUMMARY:
The purpose of this study was to determine the minimum effective dose of a local anesthetic for proper anesthesia for popliteal sciatic nerve block under ultrasound guidance in patients undergoing surgery for diabetic foot disease.

DETAILED DESCRIPTION:
Unlike general patients, patients with diabetic foot disease often have diabetic neuropathy and thus have increased sensitivity to local anesthetics. Therefore, when performing sciatic nerve block, it is essential to properly adjust the dose to prevent neurotoxicity and delay in recovery due to local anesthetics.

If the appropriate effective dose of local anesthetic for sciatic nerve block is found in patients with diabetic foot through this study, it is expected that it will be a useful basis for establishing a safe anesthetic method in the case of diabetic foot surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who can be operated under popliteal sciatic nerve block among patients undergoing surgery for diabetic foot disease

Exclusion Criteria:

1. Infection of the popliteal region
2. Severe coagulation abnormality
3. Allergic reaction or hypersensitivity to local anesthetics
4. Neurological abnormalities other than diabetic neuropathy in the lower extremity of the operation site
5. When it is impossible to evaluate sensory blockage and motor blockage
6. When the patient refuses

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Median effective anesthetic concentration 90 (MEAC 90) | within 30 minutes from the popliteal sciatic block
  Concentration of ropivacaine required for successful sciatic nerve block in 90% of all patients

SECONDARY OUTCOMES:
Median effective anesthetic concentration 50 (MEAC 50) | within 30 minutes from the popliteal sciatic block
  Concentration of ropivacaine required for successful sciatic nerve block in 50% of all patients
Sensory block onset time | within 30 minutes from the popliteal sciatic block
  Check for sensory blockade every 5 minutes until 30 minutes after block performed. For sensory block, cold sense using alcohol swabs is evaluated on the foot, comparing with the opposite foot, on a 3-point scale (0 points if there is no cold sense at all, 1 point if there is a decrease, 2 points if it is the same with the opposite foot).
  The time it takes to block to 0 point is the sensory blockade onset time.
Motor block onset time | within 30 minutes from the popliteal sciatic block
  Check for motor blockade every 5 minutes until 30 minutes after block performed. Dorsiflexion and plantar flexion is evaluated, compared to the opposite foot, on a 3-point scale (0 points for inability to move 1 point for reduced movement 2 points for normal movement).
  The time it takes to block to 0 point is the motor blockade onset time.
Block duration | within 24 hours post-operatively
  Block duration is the time from when block is performed until the patient first complained of pain at the surgical site post-operatively.
Time to first rescue analgesia | within 24 hours post-operatively
  Time to first rescue analgesia is the time from when block is performed until the patient first requested of rescue analgesics post-operatively.
Any adverse events | within 24 hours post-operatively
  Unintentional nerve damage that occurs during nerve block, pain, bleeding, infection, hypoxia, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Seokha Yoo, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea